CLINICAL TRIAL: NCT03285659
Title: Study Protocol: Development and Assessment of an Active Strategy for the Implementation of a Collaborative Care Approach for Depression in Primary Care. The INDI·i Project
Brief Title: Development and Assessment of the Implementation of a Collaborative Care Approach for Depression in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P17/077
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Depression
Keywords: depression; Primary Health Care; Health Plan Implementation; Collaborative care; Patient-Centered Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: INDI Implementation (Experimental): Primary care centres which will implement the collaborative (INDI) care model for depression
  Interventions: Other: Intervention: INDI Implementation
- Control: no INDI implementation (No Intervention): Primary care centres in which the collaborative care strategy INDI will not be implemented, but will be compared in terms of their clinical practice towards depression

INTERVENTIONS:
Other: Intervention: INDI Implementation — Implementation of a collaborative care model in the context of primary care to manage depression
  Other Names: INDI
  Arms: Intervention: INDI Implementation

SUMMARY:
Depression is one of the most common conditions among primary care patients. Nevertheless, there are several problems in depression diagnosis, clinical management and outcomes. The INDI study, which is based in a collaborative care model, aims to improve the management of depression in primary care patients. It is intended to be implemented in clinical practice within the context of primary care.

DETAILED DESCRIPTION:
BACKGROUND Depression is one of the most common conditions among primary care patients. Nevertheless, there are several problems in its diagnosis, clinical management and outcomes. The INDI study, which is based in a collaborative care model, aims to improve the management of depression in primary care patients. INDI has been proved previously to be an efficient intervention showing clinical and socio-economic benefits. INDI is intended to be implemented in the clinical practice within the context of primary care.

METHOD Aim: Test the feasibility and the impact of an implementation strategy of the INDI model for the management of depression in primary care.

Design: This is a casi-experimental study within the context of primary care. Specific geographic areas will be identified to implement the INDI program (intervention group) and other areas with similar features will to be compared (control group.

Participants: Patients diagnosed with depression will be invited to voluntarily participate in this study. Additionally, the investigators will also consider as participants the health professionals, the centres of primary care, as well as the health organizations of the geographic areas where the study will take place: Camp de Tarragona and Valles Occidental (Catalonia, Spain).

Intervention: The INDI model is a health care program for improving the management of depression. INDI includes clinical, training and organizational interventions with the participation of nurses as care managers. An active strategy based on the Promoting Action on Research Implementation in Health Services's model (PARIHS) will be designed for the implementation.

Evaluation: This study will use qualitative and quantitative methods to obtain data on the variables related to a successful implementation: feasibility, acceptability, and impact.

Discussion: In this study, the investigators aim to test the feasibility of a clinical intervention INDI, based on a collaborative care model, in the management of depression in primary care setting. If the implementation of such intervention is successful, then the achieved data and experience will help to plan a strategy to generalize the INDI model to the Catalan health system. The investigators expect significant clinical benefits to the patients, the health system and to the society.

ELIGIBILITY:
Inclusion Criteria:

* Patients: adult patients with a new diagnosis of depression or a new episode of antidepressant treatment. The comorbidity of depression with other common mental disorders such as anxiety disorders or somatization disorders is not an exclusion criterion.
* Organization: Health centres (i.e. Primary care centres) of Catalonia, which are comparable in terms of their sociodemographic, healthy and organizational features

Exclusion Criteria:

* Patients: adult patients with a diagnosis of psychotic or bipolar disorder, drug or alcohol use disorder, dementia, intellectual disability, postpartum depression, and patients included in the home care program
* Organization: no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
degree of implementation and capacity for change of the collaborative care model (INDI) | 12 months
  degree of implementation of the collaborative care model (INDI) in health organization and professionals using the Assessment of Readiness for Chronicity in Health Care Organizations (ARCHO)
patient experience about the collaborative care model (INDI) | 12 months
  how patients experience depression care according to the collaborative care model (INDI) using the Instrument for Evaluating Patient Experience of Chronic Illness Care (IEXPAC) scale

CONTACTS AND LOCATIONS:
Overall Officials: Enric Aragonès, PhD, Principal Investigator — Jordi Gol Fundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aragones E, Pinol JL, Labad A, Masdeu RM, Pino M, Cervera J. Prevalence and determinants of depressive disorders in primary care practice in Spain. Int J Psychiatry Med. 2004;34(1):21-35. doi: 10.2190/C25N-W4NY-BN8W-TXN2. PMID 15242139
- [Background] Aragones E, Pinol JL, Caballero A, Lopez-Cortacans G, Casaus P, Hernandez JM, Badia W, Folch S. Effectiveness of a multi-component programme for managing depression in primary care: a cluster randomized trial. The INDI project. J Affect Disord. 2012 Dec 15;142(1-3):297-305. doi: 10.1016/j.jad.2012.05.020. Epub 2012 Oct 11. PMID 23062747
- [Background] Aragones E, Caballero A, Pinol JL, Lopez-Cortacans G. Persistence in the long term of the effects of a collaborative care programme for depression in primary care. J Affect Disord. 2014 Sep;166:36-40. doi: 10.1016/j.jad.2014.05.003. Epub 2014 May 11. PMID 25012408
- [Background] Aragones E, Caballero A, Pinol JL, Lopez-Cortacans G, Badia W, Hernandez JM, Casaus P, Folch S, Basora J, Labad A; INDI research group. Assessment of an enhanced program for depression management in primary care: a cluster randomized controlled trial. The INDI project (Interventions for Depression Improvement). BMC Public Health. 2007 Sep 20;7:253. doi: 10.1186/1471-2458-7-253. PMID 17883845
- [Background] Aragones E, Lopez-Cortacans G, Sanchez-Iriso E, Pinol JL, Caballero A, Salvador-Carulla L, Cabases J. Cost-effectiveness analysis of a collaborative care programme for depression in primary care. J Affect Disord. 2014 Apr;159:85-93. doi: 10.1016/j.jad.2014.01.021. Epub 2014 Feb 13. PMID 24679395
- [Background] Aragones E, Comin E, Cavero M, Perez V, Molina C, Palao D. [A computerised clinical decision-support system for the management of depression in Primary Care]. Aten Primaria. 2017 Jun-Jul;49(6):359-367. doi: 10.1016/j.aprim.2016.09.011. Epub 2017 Jan 9. Spanish. PMID 28081896
- [Background] Aragones E, Pinol JL, Labad A. Depression and physical comorbidity in primary care. J Psychosom Res. 2007 Aug;63(2):107-11. doi: 10.1016/j.jpsychores.2007.05.008. PMID 17662745
- [Background] Solberg LI, Crain AL, Jaeckels N, Ohnsorg KA, Margolis KL, Beck A, Whitebird RR, Rossom RC, Crabtree BF, Van de Ven AH. The DIAMOND initiative: implementing collaborative care for depression in 75 primary care clinics. Implement Sci. 2013 Nov 16;8:135. doi: 10.1186/1748-5908-8-135. PMID 24238225
- [Background] Sighinolfi C, Nespeca C, Menchetti M, Levantesi P, Belvederi Murri M, Berardi D. Collaborative care for depression in European countries: a systematic review and meta-analysis. J Psychosom Res. 2014 Oct;77(4):247-63. doi: 10.1016/j.jpsychores.2014.08.006. Epub 2014 Aug 27. PMID 25201482
- [Background] Eccles MP, Armstrong D, Baker R, Cleary K, Davies H, Davies S, Glasziou P, Ilott I, Kinmonth AL, Leng G, Logan S, Marteau T, Michie S, Rogers H, Rycroft-Malone J, Sibbald B. An implementation research agenda. Implement Sci. 2009 Apr 7;4:18. doi: 10.1186/1748-5908-4-18. PMID 19351400
- [Background] Stetler CB, Damschroder LJ, Helfrich CD, Hagedorn HJ. A Guide for applying a revised version of the PARIHS framework for implementation. Implement Sci. 2011 Aug 30;6:99. doi: 10.1186/1748-5908-6-99. PMID 21878092
- [Background] Nuno-Solinis R, Fernandez-Cano P, Mira-Solves JJ, Toro-Polanco N, Carlos Contel J, Guilabert Mora M, Solas O. [Development of an instrument for the assessment of chronic care models]. Gac Sanit. 2013 Mar-Apr;27(2):128-34. doi: 10.1016/j.gaceta.2012.05.012. Epub 2012 Jul 24. Spanish. PMID 22832167
- [Background] Solberg LI, Asche SE, Margolis KL, Whitebird RR. Measuring an organization's ability to manage change: the change process capability questionnaire and its use for improving depression care. Am J Med Qual. 2008 May-Jun;23(3):193-200. doi: 10.1177/1062860608314942. PMID 18539980
- [Background] Kitzinger J. Qualitative research. Introducing focus groups. BMJ. 1995 Jul 29;311(7000):299-302. doi: 10.1136/bmj.311.7000.299. PMID 7633241
- [Background] Mira JJ, Nuno-Solinis R, Guilabert-Mora M, Solas-Gaspar O, Fernandez-Cano P, Gonzalez-Mestre MA, Contel JC, Del Rio-Camara M. Development and Validation of an Instrument for Assessing Patient Experience of Chronic Illness Care. Int J Integr Care. 2016 Aug 31;16(3):13. doi: 10.5334/ijic.2443. PMID 28435422
- [Background] Glasgow RE, Wagner EH, Schaefer J, Mahoney LD, Reid RJ, Greene SM. Development and validation of the Patient Assessment of Chronic Illness Care (PACIC). Med Care. 2005 May;43(5):436-44. doi: 10.1097/01.mlr.0000160375.47920.8c. PMID 15838407
- [Background] Rossom RC, Solberg LI, Vazquez-Benitez G, Crain AL, Beck A, Whitebird R, Glasgow RE. The effects of patient-centered depression care on patient satisfaction and depression remission. Fam Pract. 2016 Dec;33(6):649-655. doi: 10.1093/fampra/cmw068. Epub 2016 Aug 17. PMID 27535330
- [Background] Bolibar B, Fina Aviles F, Morros R, Garcia-Gil Mdel M, Hermosilla E, Ramos R, Rosell M, Rodriguez J, Medina M, Calero S, Prieto-Alhambra D; Grupo SIDIAP. [SIDIAP database: electronic clinical records in primary care as a source of information for epidemiologic research]. Med Clin (Barc). 2012 May 19;138(14):617-21. doi: 10.1016/j.medcli.2012.01.020. Epub 2012 Mar 22. No abstract available. Spanish. PMID 22444996
- [Background] Murray E, Treweek S, Pope C, MacFarlane A, Ballini L, Dowrick C, Finch T, Kennedy A, Mair F, O'Donnell C, Ong BN, Rapley T, Rogers A, May C. Normalisation process theory: a framework for developing, evaluating and implementing complex interventions. BMC Med. 2010 Oct 20;8:63. doi: 10.1186/1741-7015-8-63. PMID 20961442
- [Background] Serrano-Blanco A, Palao DJ, Luciano JV, Pinto-Meza A, Lujan L, Fernandez A, Roura P, Bertsch J, Mercader M, Haro JM. Prevalence of mental disorders in primary care: results from the diagnosis and treatment of mental disorders in primary care study (DASMAP). Soc Psychiatry Psychiatr Epidemiol. 2010 Feb;45(2):201-10. doi: 10.1007/s00127-009-0056-y. Epub 2009 May 19. PMID 19452110
- [Background] Gili M, Comas A, Garcia-Garcia M, Monzon S, Antoni SB, Roca M. Comorbidity between common mental disorders and chronic somatic diseases in primary care patients. Gen Hosp Psychiatry. 2010 May-Jun;32(3):240-5. doi: 10.1016/j.genhosppsych.2010.01.013. Epub 2010 Mar 1. PMID 20430226
- [Background] Community Preventive Services Task Force. Recommendation from the community preventive services task force for use of collaborative care for the management of depressive disorders. Am J Prev Med. 2012 May;42(5):521-4. doi: 10.1016/j.amepre.2012.01.010. PMID 22516494
- [Background] Thota AB, Sipe TA, Byard GJ, Zometa CS, Hahn RA, McKnight-Eily LR, Chapman DP, Abraido-Lanza AF, Pearson JL, Anderson CW, Gelenberg AJ, Hennessy KD, Duffy FF, Vernon-Smiley ME, Nease DE Jr, Williams SP; Community Preventive Services Task Force. Collaborative care to improve the management of depressive disorders: a community guide systematic review and meta-analysis. Am J Prev Med. 2012 May;42(5):525-38. doi: 10.1016/j.amepre.2012.01.019. PMID 22516495
- [Background] Coventry PA, Hudson JL, Kontopantelis E, Archer J, Richards DA, Gilbody S, Lovell K, Dickens C, Gask L, Waheed W, Bower P. Characteristics of effective collaborative care for treatment of depression: a systematic review and meta-regression of 74 randomised controlled trials. PLoS One. 2014 Sep 29;9(9):e108114. doi: 10.1371/journal.pone.0108114. eCollection 2014. PMID 25264616
- [Background] Gilbody S, Bower P, Fletcher J, Richards D, Sutton AJ. Collaborative care for depression: a cumulative meta-analysis and review of longer-term outcomes. Arch Intern Med. 2006 Nov 27;166(21):2314-21. doi: 10.1001/archinte.166.21.2314. PMID 17130383
- [Background] Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ. 2004 Nov;82(11):858-66. Epub 2004 Dec 14. PMID 15640922
- [Background] Pinto-Meza A, Fernandez A, Serrano-Blanco A, Haro JM. Adequacy of antidepressant treatment in Spanish primary care: a naturalistic six-month follow-up study. Psychiatr Serv. 2008 Jan;59(1):78-83. doi: 10.1176/ps.2008.59.1.78. PMID 18182543
- [Background] Wittchen HU, Holsboer F, Jacobi F. Met and unmet needs in the management of depressive disorder in the community and primary care: the size and breadth of the problem. J Clin Psychiatry. 2001;62 Suppl 26:23-8. PMID 11775090
- [Background] Fernandez A, Pinto-Meza A, Bellon JA, Roura-Poch P, Haro JM, Autonell J, Palao DJ, Penarrubia MT, Fernandez R, Blanco E, Luciano JV, Serrano-Blanco A. Is major depression adequately diagnosed and treated by general practitioners? Results from an epidemiological study. Gen Hosp Psychiatry. 2010 Mar-Apr;32(2):201-9. doi: 10.1016/j.genhosppsych.2009.11.015. Epub 2010 Jan 12. PMID 20302995
- [Background] Salvador-Carulla L, Bendeck M, Fernandez A, Alberti C, Sabes-Figuera R, Molina C, Knapp M. Costs of depression in Catalonia (Spain). J Affect Disord. 2011 Jul;132(1-2):130-8. doi: 10.1016/j.jad.2011.02.019. Epub 2011 Mar 12. PMID 21402411
- [Background] Sabes-Figuera R, Knapp M, Bendeck M, Mompart-Penina A, Salvador-Carulla L. The local burden of emotional disorders. An analysis based on a large health survey in Catalonia (Spain). Gac Sanit. 2012 Jan-Feb;26(1):24-9. doi: 10.1016/j.gaceta.2011.05.019. Epub 2011 Nov 9. PMID 22078690
- [Background] Gabilondo A, Rojas-Farreras S, Vilagut G, Haro JM, Fernandez A, Pinto-Meza A, Alonso J. Epidemiology of major depressive episode in a southern European country: results from the ESEMeD-Spain project. J Affect Disord. 2010 Jan;120(1-3):76-85. doi: 10.1016/j.jad.2009.04.016. PMID 19428121
- [Derived] Aragones E, Lopez-Cortacans G, Cardoner N, Tome-Pires C, Porta-Casteras D, Palao D; INDI.I Research Team. Barriers, facilitators, and proposals for improvement in the implementation of a collaborative care program for depression: a qualitative study of primary care physicians and nurses. BMC Health Serv Res. 2022 Apr 5;22(1):446. doi: 10.1186/s12913-022-07872-z. PMID 35382822
- [Derived] Aragones E, Palao D, Lopez-Cortacans G, Caballero A, Cardoner N, Casaus P, Cavero M, Monreal JA, Perez-Sola V, Cirera M, Loren M, Bellerino E, Tome-Pires C, Palacios L. Development and assessment of an active strategy for the implementation of a collaborative care approach for depression in primary care (the INDI.i project). BMC Health Serv Res. 2017 Dec 13;17(1):821. doi: 10.1186/s12913-017-2774-2. PMID 29237444